CLINICAL TRIAL: NCT06741930
Title: Potential Pro-Convulsive Properties of Ketamine and Its Effects on EEG During Procedural Sedation: A Comparative Evaluation With Midazolam and Propofol
Brief Title: Pro-Epileptic Effects of IV Ketamine
Acronym: Ketamin stdy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 35-2024
Record Dates: First submitted 2024-12-18; First posted 2024-12-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Seizure
Keywords: ketamine; midazolam; propofol; epilepsy; Procedural Sedation; Pro-Convulsive Effects
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Ketamine; Midazolam; Propofol

STUDY DESIGN:
Intervention Model Description: Single center
Who Masked: Participant, Outcomes Assessor
Masking Description: In this double-blind study, participants were randomly assigned to one of the three treatment groups (Ketamine, Midazolam, or Propofol) using a sealed envelope randomization. Both the physicians who assessed the results and the patients were blinded to the assigned group. Each participant was assigned an identification number indicating the treatment group. An emergency nurse prepared the treatment solutions immediately before administration, based on the assigned identification number, and stored them in labeled containers with no indication of their contents. A clinician with 32 years of experience, who was blinded to the study's null hypothesis and did not participate in the evaluation of results, administered the treatments and recorded patient data onto a predesigned case data form. Another physician with 27 years of experience, who was not present during the treatment, assessed the EEG recordings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketamine group (Active Comparator): The Ketamine group received IV ketamine at a dosage of 0.5-1.0 mg/kg.
  Interventions: Drug: Ketamine
- Midazolam group (Active Comparator): The Midazolam group received IV midazolam at a dosage of 0.15-0.40 mg/kg.
  Interventions: Drug: Midazolam
- Propofol group (Active Comparator): The Propofol group received IV propofol at a dosage of 0.5-1.0 mg/kg.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — The Ketamine group received IV ketamine at a titrated dose of 0.5-1.0 mg/kg with IV fentanyl, administered in small incremental boluses of 25-50 mcg to ensure adequate analgesia.
  Arms: Ketamine group
Drug: Midazolam — The Midazolam group received IV midazolam at a titrated dose of 0.15-0.40 mg/kg with IV fentanyl, administered in small incremental boluses of 25-50 mcg to ensure adequate analgesia.
  Arms: Midazolam group
Drug: Propofol — The Propofol group received IV propofol at a titrated dose of 0.5-1.0 mg/kg with IV fentanyl, administered in small incremental boluses of 25-50 mcg to ensure adequate analgesia.
  Arms: Propofol group

SUMMARY:
The investigators evaluated the safety and potential pro-epileptic effects of intravenous (IV) ketamine during procedural sedation in comparison with IV midazolam and IV propofol. Specifically, the study hypothesizes that IV ketamine, at doses used for procedural sedation, exhibits pro-convulsive properties, lowers the epileptic seizure threshold, and may induce interictal epileptiform discharges and/or seizures. Additionally, the investigators assessed the effects of these sedative agents on electroencephalographic (EEG) activity during procedural sedation.

DETAILED DESCRIPTION:
Patients were randomly assigned to one of three groups: the first group received IV ketamine at a titrated dose of 0.5-1.0 mg/kg, the second group received IV midazolam at a titrated dose of 0.15-0.40 mg/kg, and the third group received IV propofol at a titrated dose of 0.5-1.0 mg/kg. Procedural sedation in all groups was supplemented with IV fentanyl, administered in small incremental boluses of 25-50 mcg to ensure adequate analgesia. Baseline EEG recordings were obtained for all patients prior to the procedure. During the procedure, EEG recordings, vital parameters-including blood pressure, heart rate, and respiratory rate-and the depth of sedation were continuously monitored for all participants. The Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale was used to evaluate the depth of sedation.

The MOAA/S scale was applied as follows:

Score 5: Alert; responds readily to name spoken in a normal tone. Score 4: Mild sedation; lethargic response to name spoken in a normal tone. Score 3: Moderate sedation; responds only after the name is spoken loudly and/or repeatedly.

Score 2: Deep sedation; responds only after mild prodding or shaking. Score 1: Very deep sedation; unresponsive to physical stimulation. The target sedation level for patients was maintained between 2 and 3, depending on the procedural requirements. If necessary, the drug dose was carefully adjusted to increase or decrease sedation while ensuring the depth of sedation did not drop to level 1.

EEG recordings for all patients were performed. Electrodes were placed on the scalp according to the International 10-20 system, with 19 electrodes and 1 reference electrode, and the impedance of each electrode was maintained below 5 kilo-ohms. EEG recordings began with a 5-minute baseline recording during wakefulness, followed by continuous monitoring during the induction phase (administration of sedative drugs), and an additional 10-minute recording after sedation was achieved. Upon completion of the procedural intervention, EEG recordings were repeated for 10 minutes during the awakening phase and calm wakefulness.

After data collection, all EEG recordings were visually analyzed by a clinical neurophysiologist blinded to the administered drugs. EEG signals were evaluated using filters set between 0.5-70 Hz and a bipolar montage (double banana). Large-amplitude waves (>100 μV) were considered artifacts, and artifacts caused by eyelid or ocular movements were excluded from the analysis.

The recordings were analyzed for basic EEG activity, including alpha (8-12 Hz), beta (13-25 Hz), theta (4-7 Hz), delta (0.5-3.5 Hz), and gamma (25-40 Hz) rhythms, suppression-burst patterns, and their topographies. The presence of interictal epileptiform discharges, such as focal and/or generalized spike-wave, sharp wave, spike-slow wave, sharp-slow wave, and multiple spike-slow wave patterns, was noted. Additionally, clinical and/or subclinical ictal activity was documented.

Demographic data, including age, sex, comorbidities, and body weight, as well as vital parameters recorded before and during the procedure, EEG findings, and adverse effects following IV treatment, were systematically recorded.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged ≥18 years scheduled to undergo procedural sedation prior to esophagogastroduodenoscopy in the endoscopy unit were included in the study.

Exclusion Criteria:

* patients aged <18 years,
* pregnant or breastfeeding females,
* patients with a known history of epilepsy, previous status epilepticus, or neurological conditions such as head trauma, brain tumors, cerebrovascular events, meningitis, or encephalitis, as well as congenital or acquired structural brain anomalies.
* Individuals with a first-degree family history of epilepsy or who had used medications affecting the central nervous system (e.g., antidepressants, antipsychotics, sedatives, benzodiazepines, or opioids) within the previous month were also excluded.
* Patients were also excluded if they had a known allergy or hypersensitivity to the study drugs (IV ketamine, IV midazolam, IV propofol) or to adjunctive medications used for procedural sedation (e.g., IV fentanyl).
* Patients with a history of complications during anesthesia or previous surgical procedures, such as malignant hyperthermia or respiratory failure.
* Patients with significant movement disorders, agitation, scalp lesions, or other conditions interfering with EEG recording.
* Patients with severe cardiovascular disease, including uncontrolled hypertension, advanced heart failure, or arrhythmias, as well as those with oxygen saturation <90%, a high risk of respiratory depression, or severe obstructive sleep apnea syndrome.
* Patients with severe hepatic or renal failure, or those who had undergone major surgery within the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Rates of interictal epileptiform discharges on EEG | 0, 5, and 30 min following the initial administration.
  The investigators assessed the rates of interictal epileptiform discharges on EEG, including focal and/or generalized spike-wave, sharp wave, spike-slow wave, and sharp-slow wave patterns, induced by IV ketamine.
Rates of interictal epileptiform discharges on EEG | 0, 5, and 30 min following the initial administration.
  The investigators assessed the rates of interictal epileptiform discharges on EEG, including focal and/or generalized spike-wave, sharp wave, spike-slow wave, and sharp-slow wave patterns, induced by IV midazolam.
Rates of interictal epileptiform discharges on EEG | 0, 5, and 30 min following the initial administration.
  The investigators assessed the rates of interictal epileptiform discharges on EEG, including focal and/or generalized spike-wave, sharp wave, spike-slow wave, and sharp-slow wave patterns, induced by IV propofol.

SECONDARY OUTCOMES:
Presence of subclinical seizure activity | 0, 5, and 30 min following the initial administration.
  The investigators assessed the presence of subclinical seizure activity (ictal activity) on EEG within the ketamine group.
Presence of subclinical seizure activity | 0, 5, and 30 min following the initial administration.
  The investigators assessed the presence of subclinical seizure activity (ictal activity) on EEG within the midazolam group.
Presence of subclinical seizure activity | 0, 5, and 30 min following the initial administration.
  The investigators assessed the presence of subclinical seizure activity (ictal activity) on EEG within the propofol group.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Az A, Dogan Y. Unexpected consequences: A case of ketamine-induced seizure in procedural sedation. Turk J Emerg Med. 2024 Oct 1;24(4):259-261. doi: 10.4103/tjem.tjem_67_24. eCollection 2024 Oct-Dec. PMID 39564442
- [Result] Kim JH, Lee CK, Yu SH, Min BD, Chung CE, Kim DC. Ketamine-induced generalized convulsive seizure during procedural sedation. Arch Craniofac Surg. 2021 Apr;22(2):119-121. doi: 10.7181/acfs.2021.00094. Epub 2021 Apr 20. PMID 33957739
- [Result] Shehata IM, Kohaf NA, ElSayed MW, Latifi K, Aboutaleb AM, Kaye AD. Ketamine: Pro or antiepileptic agent? A systematic review. Heliyon. 2024 Jan 10;10(2):e24433. doi: 10.1016/j.heliyon.2024.e24433. eCollection 2024 Jan 30. PMID 38293492
- [Result] Besha A, Adamu Y, Mulugeta H, Zemedkun A, Destaw B. Evidence-based guideline on management of status epilepticus in adult intensive care unit in resource-limited settings: a review article. Ann Med Surg (Lond). 2023 Apr 17;85(6):2714-2720. doi: 10.1097/MS9.0000000000000625. eCollection 2023 Jun. PMID 37363462
- [Result] Cohen SP, Bhatia A, Buvanendran A, Schwenk ES, Wasan AD, Hurley RW, Viscusi ER, Narouze S, Davis FN, Ritchie EC, Lubenow TR, Hooten WM. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):521-546. doi: 10.1097/AAP.0000000000000808. PMID 29870458
- [Result] Zanos P, Moaddel R, Morris PJ, Riggs LM, Highland JN, Georgiou P, Pereira EFR, Albuquerque EX, Thomas CJ, Zarate CA Jr, Gould TD. Ketamine and Ketamine Metabolite Pharmacology: Insights into Therapeutic Mechanisms. Pharmacol Rev. 2018 Jul;70(3):621-660. doi: 10.1124/pr.117.015198. PMID 29945898